CLINICAL TRIAL: NCT05561413
Title: Randomised Controlled Feasibility Trial Evaluating the Effectiveness of Mindfulness Compared to Exercise and Mindfulness on Fatigue in Women With Gynaecology Cancer
Brief Title: Gynaecology Exercise and Mindfulness Study
Acronym: GEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/21/00 76
Record Dates: First submitted 2022-09-20; First posted 2022-09-30 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Gynecologic Cancer; Uterus Cancer; Ovary Cancer; Cervical Cancer; Vaginal Cancer; Vulvar Cancer
Keywords: Neoplasms; Mindfulness; Online
MeSH Terms: conditions — Uterine Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Neoplasms | interventions — Mindfulness; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness and exercise (Experimental): This group will undertake exercise and mindfulness for 8 weeks. The home based walking and strengthening intervention is individually tailored for each participant. All exercise demonstrations, information, reporting of activity and setting of goals will take place in the app that participants will download. Additionally this group will receive a hard copy of the goal setting diary. All mindfulness information and practices are available in the app. New content will be released each week as the participants progress through the program. Participants will be phoned weekly over the 8 weeks to monitor progress.
  Interventions: Behavioral: Mindfulness and exercise
- Mindfulness (Active Comparator): This group will undertake mindfulness only over 8 weeks. The mindfulness program is based on mindfulness-based stress reduction (MBSR). All information, practices and logging of the mindfulness practice will be done via the app that participants will download. Participants will be phoned weekly over the 8 weeks to monitor progress. New content will be released each week as participants progress through the program.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness and exercise — The mindfulness and exercise group aims to gradually increase participants exercise levels so that they begin to achieve the recommended levels along with the strengthening exercises for all major muscle groups. Along side this mindfulness will be introduced and built on to help consolidate exercise uptake and help manage symptoms experienced by the participants.
  Arms: Mindfulness and exercise
Behavioral: Mindfulness — The delivery of this practice will be through the app downloaded by participants. The practice based on mindfulness based stress reduction (MBSR). Will build on practice over the 8 weeks.
  Arms: Mindfulness

SUMMARY:
The aim of this study is to explore the feasibility and effectiveness of conducting a mindfulness and home-based walking and strength training program on fatigue, psychological outcomes and quality of life for gynecological cancer survivors. The intervention consists of a 8 week mindfulness and home based walking and strengthening program for gynecology survivors. It will be delivered through a specifically designed app. The aim would be to gradually increase exercise and mindfulness levels so participants start to achieve the recommended levels of activity per week.

Participants will be recruited via cancer Charites and their service users either directly and through social media (Facebook, Instagram, Twitter). Both groups will receive an intervention either mindfulness alone or mindfulness and exercise. Assessments will be taken at baseline (0 weeks) and post intervention (8 weeks). Both groups will complete the same assessments at the same time-points.

DETAILED DESCRIPTION:
Treatment modalities can be effective in managing and treating gynecology cancers but may lead to unwanted long term side effects. Some of which include fatigue, changes in mood and sleep disturbance. All of which can have an effect on quality of life. Both exercise and mindfulness would appear to show a positive effect on managing some of these symptoms. However, not only does ambiguity continue around the effect of these interventions on symptoms of cancer but continues to be a lack of evidence for certain types of cancer such as gynecology. Furthermore, combining interventions that individually are effective may enhance effectiveness when used together and the delivering these online may reach a wider population. The evidence for this is also lacking within the literature. Therefore this study aims to assess the feasibility of delivering these interventions through an online platform to assess not only the acceptability but also effect on clinical outcomes.

Participants will be recruited through contact via cancer charities and online (Social media), they will self refer to the team and will be assessed for eligibility. If eligible and interested participant information sheet will be sent electronically and time given (one week) to consider study. Contact will be made with participant after this time and if interested a link to electronic consent will be sent. On receiving the completed consent another link will be sent to participant for completion of baseline outcome measures. The outcome measures assessed include feasibility, fatigue, physical activity level, mood (anxiety/depression), sleep, quality of life and mindfulness. Following randomization both groups will be given instructions on how to download app and reporting of activity. Both groups will be contacted through weekly phone calls to monitor their progress. Once 8 weeks have been completed a link will be sent to participants to complete the post-intervention outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I-IV gynecologic cancer including endometrial, ovarian, cervical, vaginal, vulva, fallopian tube.
* Experiencing fatigue and at screening have a numerical rating score of ≥4 on a scale of 0-10.
* Ambulatory and without the use of a walking aid.
* Currently sedentary (exercising < once a week for 20 minutes at a vigorous intensity or, two times per week for 30 minutes at moderate intensity or < 20 minutes three times per week, for the past 6 months).

Exclusion Criteria:

* Currently actively and regularly practicing mindfulness.
* Have a confirmed diagnoses of Schizophrenia spectrum disorder, Bipolar disorder, Post-traumatic stress disorder, or risk factors for psychosis (eg personality disorder)
* Have an existing medical condition that may inhibit safe participation in the exercise part of the intervention study.
* Previously diagnosed with a fatigue-related co-morbid medical condition (i.e. Fibromyalgia, Chronic Fatigue Syndrome, Multiple Sclerosis (MS), Myalgic Encephalopathy (ME), Lupus or Arthritis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants that describe themselves as female gender eligible to participate.
Enrollment: 40 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of eligibility and enrollment | 12 months
  Number of eligible participants, and the proportion of those eligible that enrolled will be assessed to evaluate the feasibility of eligibility and enrollment.
Retention rate in study as feasibility | 8 weeks
  Number and proportion of participants completing all assessments.
Feasibility as assessed by rate of attrition | 8 weeks
  The number of participants dropping out after start of intervention for any reason will be assessed to evaluate attrition rate.
Feasibility as assessed by adherence | 8 weeks
  Will be assessed by frequency and duration of practicing of exercise and mindfulness (recorded in a log via app).

SECONDARY OUTCOMES:
Fatigue | Week 0 and 8
  The Functional Assessment of Chronic Therapy- Fatigue (FACIT-F) subscale will be used a 13- item questionnaire that uses a 5 point Likert scale. The lower the score on this scale indicates the greater the fatigue with scores less than 20 representing severe fatigue and scores greater than 45 as normal.
Evaluate the Quality of Life | Week 0 and 8
  The Functional Assessment of Cancer Therapy General (FACT-G) is a 28- item rated scale. It assesses physical, social, emotional and functional wellbeing. Higher scores in this questionnaire indicate better quality of life.
Psychological outcomes | Week 0 and 8
  The psychological outcomes will be assessed using the Hospital Anxiety and Depression Scale (HADS). This questionnaire has 14 questions, 7 each for assessing anxiety and depression. A HADS score of greater than 11 is more defining of anxiety and depression, with a reduction of 3 points indicating a clinical improvement.
Sleep | Week 0 and 8
  The Pittsburgh Sleep Quality Index (PSQI) a 19 items questionnaire that measures 7 domains of sleep scored on a 0-3 scale over 1 month will be used. The questionnaire gives a score that ranges from 0-21 with the higher the score the worse the sleep quality.
Mindfulness | Week 0 and 8
  The 24 item Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) is a 5 point Likert Scale which assess mindfulness in daily life. It measures 5 sub-scales: observing, describing, acting with awareness, non-judgement of inner experience and non-reacting to inner experience. The higher the score the greater the mindfulness.
Physical activity | Week 0 and 8
  International physical activity questionnaire (IPAQ) short form will be used to evaluate the effects on levels of activity

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Gracey, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Belfast, Antrim, United Kingdom

REFERENCES:
- [Derived] McCloy K, Hughes C, Dunwoody L, Marley J, Cleland I, Cruciani F, Saunders C, Gracey J. Evaluating the effectiveness of mindfulness alone compared to exercise and mindfulness on fatigue in women with gynaecology cancer (GEMS): Protocol for a randomised feasibility trial. PLoS One. 2023 Oct 26;18(10):e0278252. doi: 10.1371/journal.pone.0278252. eCollection 2023. PMID 37883461